CLINICAL TRIAL: NCT06111339
Title: Ketamine for the Treatment for Opioid Use Disorder and Suicidal Ideation in the Emergency Department
Brief Title: Ketamine for OUD and Suicidal Ideation in the ED
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low recruitment numbers and study funding will be closing shortly.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Director, Division of Addiction Psychiatry, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023P002857
Record Dates: First submitted 2023-10-19; First posted 2023-11-01 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Opioid Use Disorder; Suicidal Ideation
MeSH Terms: conditions — Opioid-Related Disorders; Suicidal Ideation | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will then be randomized in a double-blind fashion to receive either ketamine (0.8 mg/kg) or a matched volume saline placebo in the ED. Randomization will use a permuted block method58. The randomization ratio will be 1:1. A biostatistician will generate the randomization codes and provide the randomization list to the hospital's Investigational Drug Services (IDS). The study RA will contact IDS once the participant has signed informed consent and IDS staff will randomize participants. Both RA, study team and the clinical team will be blinded to the allocation.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): This arm will receive ketamine (n=25)
  Interventions: Drug: Ketamine
- Saline Placebo (Placebo Comparator): This arm will receive the saline placebo (n=25)
  Interventions: Other: Saline Solution

INTERVENTIONS:
Drug: Ketamine — The intervention will consist of a single infusion of ketamine in the ED at a dose of 0.8mg/kg over 40 minutes.
  Arms: Ketamine
Other: Saline Solution — The placebo will be a 0.9% saline solution administered over 40 minutes.
  Arms: Saline Placebo

SUMMARY:
This is a pilot, double-blind, placebo-controlled randomized clinical trial of individuals with opioid use disorder (OUD) with suicidal ideation in the emergency department (ED) to receive either a single infusion of ketamine 0.8mg/kg (n=25) or saline placebo (n=25). The primary aim is to evaluate the safety of the ketamine treatment. The secondary aim is to determine the preliminary efficacy of opioid- and suicide-related outcomes.

DETAILED DESCRIPTION:
Individuals with opioid use disorder (OUD) seeking medical care in the emergency department (ED) will be first evaluated as per usual clinical care by the ED staff, including any acute medical treatment for overdose or any other acute medical issues needing treatment. For those who endorse suicidal ideation, after medical clearance, the standard medical care will involve the evaluation of patients by the psychiatry consult service in the ED. Patients evaluated by psychiatry who require further behavioral health care and do not have acute medical issues remain in the ED awaiting admission to an inpatient psychiatry unit or other linkages to care. Potential participants will be approached after the psychiatry evaluation is complete and a decision has been made to keep the patients in the ED for continued psychiatric care or admit them medically. After applying the full inclusion and exclusion criteria, those who remain eligible will be randomized to receive in a double-blind fashion either a single infusion of ketamine (0.8mg/kg) or a saline placebo. Safety assessments will be conducted during and after the receipt of ketamine or placebo, and at follow-up assessments after discharge from the emergency department of the hospital following inpatient psychiatric treatment.

ELIGIBILITY:
Inclusion/Exclusion Criteria:

To be eligible, individuals must be/have:

* English speaking adults aged 18 and above
* Diagnosed with DSM5 opioid use disorder, moderate or severe, or clinically suspected opioid use disorder
* Endorsing suicidal ideation sufficiently severe to meet criteria for referral to an inpatient psychiatric facility or a crisis stabilization unit
* Any prior history of an opioid overdose
* Medically cleared

Individuals with any of the following will be excluded:

* Any psychotic disorder or active homicidally
* Inability to perform consent due to impaired mental status
* Current substance intoxication or current (or within the past 1-month) mania, hypomania, mixed-episode, or psychosis
* Systolic blood pressure persistently elevated above 160mmHg, diastolic blood pressure greater than 100 mmHg, or heart rate >100bmp, in the ED
* Clinical Opioid Withdrawal Scale (COWS) score of 12 or greater
* History of hypersensitivity to ketamine, or experience of emergence reaction
* History of hypersensitivity to ondansetron or concurrently using apomorphine
* History of any illicit or recreational use of ketamine in the past 12 months
* Receipt of ketamine treatment for depression in the past 3 months
* History of DSM5 hallucinogen use disorder, intracranial mass or bleed, porphyria, thyrotoxicosis, seizure disorder other than from alcohol withdrawal, liver cirrhosis, or sleep apnea
* Cardiac or EKG abnormalities based on history, physical examination or the baseline EKG
* History within 6 months of thoracic surgery, lung cancer, head trauma, stroke, or myocardial infarction
* Liver dysfunction with LFTs >3x upper normal limit
* Current use of medications with known drug-drug interactions with ketamine (i.e., St. John's Wort, theophylline, opioid analgesics other than buprenorphine and methadone for the treatment OUD, Central Nervous System (CNS) depressants other than benzodiazepines or phenobarbital)
* Pregnant
* Patients who are breastfeeding
* ASA class 3 or greater or documented history of difficult airway in HER
* Active exacerbation of COPD or asthma
* Currently participating or anticipated to participate in a concurrent investigational clinical trial
* High risk for adverse emotional or behavioral reaction based on the opinion of the study investigators, including evidence of a personality disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2024-06-14 (Actual); Primary Completion 2025-03-11 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Lower Suicidal Ideation | 7-day remote follow up; 14- day remote follow up; 28 days after being discharged from inpatient unit or emergency department.
  For suicidal ideation, the Columbia Suicide Severity Rating Scale (C-SSRS), which is a 5-item tool, will be used to assess suicidal ideation.
Less Illicit Opioid Use | 28 days after being discharged from inpatient unit or emergency department.
  For illicit opioid use, the outcome is the proportion of abstinent days during the 28-day period after discharge from the ED or the inpatient psychiatric unit, assessed using the self-report Timeline Follow Back (TLFB). The TLFB is a gold-standard calendar method to assess substance use in the prior 28 days.
Incidence of Serious Adverse Events (SAE) | From the beginning on the infusion, every 15 minutes throughout infusion, and at the end of the infusion.
  The primary safety outcome is the incidence of serious adverse events (SAE) defined as hypertensive urgency (SBP>180mmHg or DBP>110mmHg) or tachycardia (HR>130bmp). Vital signs will be monitored throughout the ketamine administration.

SECONDARY OUTCOMES:
Opioid Withdrawal | Assessed daily while the participant remains in the ED, starting with the day that the ketamine/placebo infusion occurs until the discharge date.
  Opioid withdrawal will be measured using the Clinical Opioid Withdrawal Scale (COWS). Scoring: 5-12 = mild 13-24 = moderate 25-36 = moderately severe >36 = severe withdrawal
Days to Relapse | 7-day remote follow up; 14- day remote follow up; 28 days after being discharged from inpatient unit or emergency department.
  Days to Relapse will be assessed using the self-report Timeline Follow Back (TLFB). The TLFB is a gold-standard calendar method to assess substance use in the prior 28 days.
Percentage of Addiction Treatment Engagement | 28 days after being discharged from inpatient unit or emergency department.
  Evaluating whether the patient is engaged or not in treatment, such as meeting their primary care physician or addiction specialist.
Urine Toxicology Result for Ketamine | 28 days after being discharged from inpatient unit or emergency department.
  The urine drug screen result (positive or negative) for ketamine will be assessed.
Urine Toxicology Result for Opioids | 28 days after being discharged from inpatient unit or emergency department.
  The urine drug screen result (positive or negative) for opioids will be assessed.
Emergence of Psychiatric Adverse Effects | 28 days after being discharged from inpatient unit or emergency department.
  The CADSS is a scale with 6 subject-rated items. Items are divided into 3 components-depersonalization, derealization, and amnesia.
Emergence of Psychiatric Adverse Effects | 28 days after being discharged from inpatient unit or emergency department.
  The PRISE is a patient self-report tool used to qualify side effects in the following domains: gastrointestinal, heart, skin, nervous system, eyes/ears, genital/urinary, sleep, sexual functioning, and other. Each domain has multiple symptoms which can be endorsed. For each domain the patient rates whether the symptoms are tolerable or distressing
Craving for Opioids | 7-day remote follow up; 14- day remote follow up; 28 days after being discharged from inpatient unit or emergency department.
  The Opioid Craving Questionnaire (3-item scale) will assess opioid craving. Each question assesses opioid craving with answer choices ranging from 0 (not at all) to 10 (extremely strong) or 0 (not at all) to 10 (I'm sure I would use opiates). A higher score for each question indicates higher opioid cravings.
Craving for Ketamine | 7-day remote follow up; 14- day remote follow up; 28 days after being discharged from inpatient unit or emergency department.
  The Ketamine Craving Questionnaire (3-item scale) will assess ketamine craving. Each question assesses ketamine craving with answer choices ranging from 0 (not at all) to 10 (extremely strong) or 0 (not at all) to 10 (I'm sure I would use ketamine). A higher score for each question indicates higher ketamine cravings.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States